CLINICAL TRIAL: NCT02785068
Title: A Phase 1 Study Combining MM-151 + Nal-IRI + 5-FU + Leucovorin in RAS/RAF Wild-type Metastatic Colorectal Cancer
Brief Title: Evaluation of MM-151 + Nal-IRI + 5-FU + Leucovorin in RAS/RAF Wild-type Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-151-06-12-04
Record Dates: First submitted 2016-05-11; First posted 2016-05-27 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: Phase I; Cancer; EGFR; Metastatic Colorectal Cancer; Oncology; RAS/RAF Wild-Type; Nal-IRI; EGFR Inhibitor; Oligoclonal Antibody; Nanoliposome; Nanoliposomal Irinotecan
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — MM-151; irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1b/2a (Experimental): Phase 1b: Safety Evaluation - MM-151 (weekly dosing) in combination with fixed doses of nal-IRI 70mg/m2 + Leucovorin 400 mg/m2 + 5-FU 2400mg/m2 every two weeks.
  Phase 2a: Expansion - MM-151 (Maximum Tolerated Dose or Recommended Phase 2 Dose) in combination with fixed doses of nal-IRI 70mg/m2 + Leucovorin 400 mg/m2 + 5-FU 2400 mg/m2.
  Interventions: Drug: MM-151; Drug: nal-IRI; Drug: Leucovorin; Drug: 5-FU

INTERVENTIONS:
Drug: MM-151 — Oligoclonal antibody
Drug: nal-IRI — Nanoliposomal irinotecan
  Other Names: MM-398; Onivyde
Drug: Leucovorin — folinic acid
  Other Names: folinic acid
Drug: 5-FU — Chemotherapy
  Other Names: fluorouracil

SUMMARY:
A phase 1b/2a study evaluating the combination of MM-151 + nal-IRI + 5-FU + Leucovorin in RAS/RAF wild-type Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
Part 1: Patients will be enrolled to determine the maximum tolerated dose, safety and tolerability of MM-151 + nal-IRI + 5-FU + LV in patients with mCRC that are RAS/RAF wild-type.

Part 2: Patients will be enrolled at the maximum tolerated dose of MM-151 in combination with nal-IRI + 5-FU + LV to characterize initial efficacy in conjunction with levels of irinotecan and SN-38 measured in tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than 18 years of age
* Patients must be able to provide informed consent
* Patients must have KRAS/NRAS/BRAF wild-type colorectal cancer
* Willing to abstain from sexual intercourse or to use an effective form of contraception during the study and for 120 days following the last dose of any study therapy). This applies to women of childbearing potential as well as fertile men and their partners

Exclusion Criteria:

* Patients who have had previous pelvic radiation treatment
* Patients who are pregnant or lactating
* Patients who have untreated (primary) or uncontrolled Central Nervous System (CNS) (primary or metastatic) malignancies; patients with CNS metastases who have undergone surgery or radiotherapy or who have been on a stable dose of corticosteroids for at least 2 weeks and whose disease is stable prior to the first scheduled day of dosing will be eligible for the trial.
* History of any second malignancy in the last 3 years; patients with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible.
* Patients who have received other recent antitumor therapy including any standard chemotherapy or radiation within 14 days and bevacizumab within 28 days (and having passed the time of any actual or anticipated toxicities) prior to the first scheduled dose of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
To find the phase II dose of MM-151 based on safety and tolerability of MM-151 + nal-IRI + 5-FU + Leucovorin that will be assessed through evaluation of dose limiting toxicity reporting. | The DLT timeframe is from date of first dose up until 42 days after that date
To correlate disease response according to RECIST with levels of irinotecan and SN-38 in tumor tissue | 2 years

SECONDARY OUTCOMES:
The number of participants with adverse events (AE) related to treatment with MM-151 + nal-IRI + 5-FU + leucovorin, assessed according to NCI CTCAE v4.0 | 2 years
  These will be described by abnormalities in hematology, blood chemistry and other laboratory abnormalities, ECG, physical examination, vital signs and other safety parameters.
  Frequency, duration and severity of the adverse events according to NCI CTCAE v4.0 will be assessed.
The PK parameters of MM-151 and nal-IRI will be described per Cmax | Priming Phase Day 1, Priming Phase Day 8, C1D1, C1D8, C1D15, C1D22, C2D1, C2D15, C2D17, C2D22, C3D1, C5D1
The PK parameters of MM-151 and nal-IRI will be described per AUC | Priming Phase Day 1, Priming Phase Day 8, C1D1, C1D8, C1D15, C1D22, C2D1, C2D15, C2D17, C2D22, C3D1, C5D1
Objective response based on RECIST | 2 years
Measure pre-treatment and on-treatment levels of EGFR ligands | 2 years
Presence of anti-drug antibodies will be assessed | 2 years

IPD SHARING:
Plan to Share IPD: No